CLINICAL TRIAL: NCT03095794
Title: Brain Mechanism of Social Decision-making
Brief Title: Social Decision-making (SOCIAL-DECISION)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient on-site staff to manage study
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0679
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neural mechanisms of decision making (Experimental): Previous studies on how brain manages a value-based decision have been bounded to individual decisions. The current study will extend the understanding of social dimensions by answering four questions.
  Interventions: Other: How people learn another's value preference during decision under risk; Other: Neural mechanism of making a group decision under risk that influences on in-group members; Other: Neural mechanism of making a group decision that influences on out-group members; Other: fMRI

INTERVENTIONS:
Other: How people learn another's value preference during decision under risk — The aim of this study is to investigate how an agent learns another's value preference when they should make decisions on behalf of another. This experiment consists of 3 parts(i) measuring individual's loss aversion; (ii) feedback based learning of another's value preference; (iii) and decisions on behalf of others.
Other: Neural mechanism of making a group decision under risk that influences on in-group members — how individuals evaluate the risk and the outcome when they should make a single agreement decision in a group that will influence every member's payoff regardless of individuals' decisions. For the first part of the experiment, we will measure the individual level of loss aversion which will be used as the parameter for controlling individual differences.
Other: Neural mechanism of making a group decision that influences on out-group members — Human is decimated with other species by delegation of one responsibility. Although the person who has no-interests with the outcome of decision, they should make a delegated decision. Therefore, this decision has influences on others who are not part of the group. The third party punishment (Juries decision making) is one example of the decision made by a group influencing the out group members.
Other: fMRI — For neuroimaging passes, the expected duration of each of the experimental protocols is about 1h30 for tasks 1 and 2 and about 2h for task 3. The maximum period foreseen for neuroimaging tests is 3 years and will start as soon as possible. Completion of the behavioral tests.

SUMMARY:
The purpose of this study is to investigate neural mechanism of healthy humans underlying group decision making and compare it with that of individual decision-making. Using functional neuroimaging technology combining with computational modeling, we examine how the human brain process social information to make a decision within a group, which often guides humans to make a better decision using collective wisdom.

ELIGIBILITY:
Inclusion Criteria:

* healthy human adult
* normal vision

Exclusion Criteria:

* depression
* potential addiction to alcohol/ nicotine

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2016-07-18 (Actual)

PRIMARY OUTCOMES:
Brain activation associated with decision-making (fMRI, non-invasive measure) | Day 1
  1 hour in a fMRI scanner

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEMILY, MD, Principal Investigator — CH le Vinatier
Locations (1):
- CH le Vinatier, Bron, France